CLINICAL TRIAL: NCT04987099
Title: Effects of Increased Maternal Choline Intake on Child Cognitive Development
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1911009219
Record Dates: First submitted 2021-02-18; First posted 2021-08-03 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Pregnancy
Keywords: Choline; Prenatal Supplementation; Pregnancy; Offspring Cognition; Offspring Emotion Regulation
MeSH Terms: interventions — Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only a Laboratory Manager, who will label the supplements with participant ID, will have access to participants' study assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Dose (Experimental): Participants will consume a 15 mL grape juice cocktail solution that contains 550 mg of choline once daily for the duration of their pregnancy.
  Interventions: Dietary Supplement: 550 mg/day Choline
- Control Dose (Placebo Comparator): Participants will consume a 15 mL grape juice cocktail solution that contains 25 mg of choline once daily for the duration of their pregnancy.
  Interventions: Dietary Supplement: 25 mg/day Choline

INTERVENTIONS:
Dietary Supplement: 550 mg/day Choline — Choline chloride (550 mg) is a water soluble choline salt that will be provided in a grape juice cocktail solution to participants for daily consumption.
  Arms: Experimental Dose
Dietary Supplement: 25 mg/day Choline — Choline chloride (25 mg) is a water soluble choline salt that will be provided in a grape juice cocktail solution to participants for daily consumption.
  Arms: Control Dose

SUMMARY:
The purpose of this study is to examine cognitive and affective outcomes in the offspring of women supplemented with choline vs. control during pregnancy.

DETAILED DESCRIPTION:
Choline, an essential nutrient, plays numerous important roles in fetal development. However >90% of pregnant women in the U.S. consume less than the recommended amount, and choline is typically absent from most prenatal vitamins. Moreover, current choline recommendations for pregnant women may be inadequate for optimal fetal development and lifelong health. Animal studies clearly show that maternal choline supplementation (MCS) improves offspring memory, attention, and emotion regulation. The purpose of this study is to examine cognitive and affective outcomes in the offspring of women supplemented with choline vs. control during the second and third trimesters of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Singleton pregnancy (carrying one baby)
* 21-40 years old
* Between 12-18 weeks pregnant at the time of screening
* Self-reported BMI <35.0 in the three months prior to pregnancy (estimated or known)
* Willingness to comply with all study procedures for the duration of the study
* Intending to live in Ithaca, NY or the surrounding area for the duration of the study
* Intending to deliver at Cayuga Medical Center

Exclusion Criteria:

* Self-reported history of health conditions associated with metabolic or gastrointestinal function or adverse child outcomes
* Current use of medications known to affect liver or kidney function or child outcomes
* High omega-3 fatty acid intakes from diet (as determined by a licensed registered dietitian) at screening
* Choline supplementation that exceeds 50 mg/day at screening
* Use of alcohol, tobacco products, or recreational drugs during pregnancy or during the Prenatal Phase of the study
* Use of non-study approved or provided supplements during the Prenatal Phase of the study
* Development of pregnancy-related complications during the study (i.e. gestational diabetes, gestational hypertension, preeclampsia, genetic abnormalities, or miscarriage)

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The Effects of Maternal Choline Supplementation on Infant Visual Recognition Memory: Developmental Trajectory Analysis of the Novelty Preference Score | Infant ages of 5, 7, 10, and 13 months
  The composite novelty score (proportion of looking to the novel image) is obtained from a series of 9 visual paired comparison tests. The novelty score is a measure of visual recognition memory for infants and has been shown to predict cognitive outcomes in childhood. This analysis will assess developmental trajectories for performance on this task across the first year of life (ages 5, 7, 10, and 13 months).
The Effects of Maternal Choline Supplementation on Infant Visual Attention: Mean Orienting Speed Score | Infant ages of 5, 7, 10, and 13 months
  Visual attention orienting speed is measured by the latency to initiate a stimulus-guided fixation shift to a peripheral visual target (mean of up to 20 target presentations). The orienting score is found to be sensitive to maternal choline supplementation in infants of this age and has shown acceptable test-retest reliability and prediction of attention, memory, and intelligence quotient outcomes in childhood. This analysis will assess the within-subject age-adjusted mean saccade latency obtained from tests repeated at ages 5, 7, 10, and 13 months.
The Effects of Maternal Choline Supplementation on Infant Sustained Focused Attention: Mean Sustained Focused Attention Score | Infant ages of 5, 7, 10, and 13 months
  Sustained focused attention is measured during a 5-minute period in which infants are engaged in solitary play with a complex toy. The score is the average duration of infant engagement in a state of focused attention on the toy. Infants who sustain focused attention for longer durations have been found to have fewer attentional problems as children. This analysis will assess the within-subject age-adjusted mean duration of focused attention obtained from tests repeated at ages 5, 7, 10, and 13 months.
The Effects of Maternal Choline Supplementation on Emotion Regulation: Lab-TAB/Frustation Task Scores | Infant ages of 7, 10, and 13 months
  Negative affect in response to goal blockage is measured by coding of infant facial expression, vocalization, and body language over the course of four sequential task trials to produce composite scores of negative affect. Infants' ability to regulate negative affect during the task has been found to predict aggressiveness at age three and has been associated with non-compliance in toddlerhood.
The Effects of Maternal Choline Supplementation on Emotion Regulation: Face-to-Face Still-Face Paradigm Scores | Infant ages of 7, 10, and 13 months
  Infant negative affect in response to a violation of social expectations for interactions with a parent (the parent not engaging with infant's social cues and maintaining a neutral expression) is measured by coding of infant negative vocalizations (crying, screaming, etc.) over the course of three sequential task trials to produce composite scores of negative affect. Infants' behavior in this task has been shown to predict later attachment, internalizing, and externalizing behaviors in toddlerhood and early childhood.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Strupp, PhD, Principal Investigator — Cornell University
Locations (1):
- Cornell University, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: No